CLINICAL TRIAL: NCT04909866
Title: The Efficacy and Safety of TACE, Lenvatinib and Camrelizumab in the Treatment of BCLC Stage B/C Hepatocellular Carcinoma: a Single-arm, Single-center, Open-label Study
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Bin Xiong, Principal Investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CXPJJH12000001-2020223
Record Dates: First submitted 2021-02-09; First posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE+Lenvatinib+Camrelizumab (Experimental)
  Interventions: Combination Product: TACE+Lenvatininb+Camrelizumab

INTERVENTIONS:
Combination Product: TACE+Lenvatininb+Camrelizumab — Patients included in the trial were treated with TACE, lenvatinib combined with Camrelizumab.

SUMMARY:
This study is a single-center, single-arm, open-label prospective clinical trial. By recording the disease-free progression (PFS), overall survival (OS) and tumor treatment response of the included patients, it is planned to evaluate TACE, lenvatinib and carrelizumab in the treatment of BCLC B/C hepatocytes Survival benefits of cancer patients; at the same time, the immune indicators before and after treatment are tested, the dosage is optimized, and the mechanism of combination therapy in liver cancer is explored to lay the foundation for screening more suitable treatment populations; laboratory testing indicators and adverse events To observe and evaluate the safety of combined therapy; adopt immunohistochemistry, pathology, cell biology, proteomics and imagingomics methods to comprehensively evaluate the changes after combined therapy.

DETAILED DESCRIPTION:
At present, the treatment methods for advanced liver cancer mainly include local interventional therapy, targeted therapy and immunotherapy.This study focused on patients with primary HCC diagnosed clinically and radiologically, histologically, or cytologically, in BCLC stage B/C.To study the medium and long-term efficacy of TACE and remvaritinib combined with carrelizumab in the treatment of BCLCB/C stage liver cancer, and to evaluate its effectiveness;To evaluate the safety and efficacy of remvatinib combined with carrelizumab in the treatment of liver cancer, and to clarify the application value of combined therapy, so as to lay a foundation for the evaluation of clinical efficacy in patients with middle and advanced liver cancer.Immune checkpoint inhibitors and cell-based cancer immunotherapies have been widely used in a variety of advanced malignancies by modulating the tumor immune response.Studies have shown that programmed death receptor 1 (PD-1) is an immune checkpoint molecule that negatively regulates the immune function of T cells through interaction with its ligand PD-L1.A growing body of evidence suggests that the PD-1/PD-L1 interaction is one of the major cancer avoidance mechanisms in humans.Overexpression of PD-L1 or PD-L2 by tumor cells interacts with PD-1 molecules expressed in activated T cells to inhibit T cell receptor (TCR) signal transduction, and eventually leads to inactivation of effector T cells and loss of proliferative ability, leading to tumor immune escape.Based on this mechanism of tumors, new immunotherapies that block the interaction between PD1/PD-L1 have been produced, changing the treatment strategies of various malignant tumors.By inhibiting the negative regulatory effect of PD-1/PD-L1 pathway on T cells, the anti-tumor immune response of the body can be enhanced, the T cell response activity targeting the patient's tumor can be improved, and the proliferation of effector T lymphocytes can be promoted, finally providing an important and lasting immune response against the patient's malignant tumor.Carrelizumab is a human high-affinity IgG4 anti-PD-1 monoclonal antibody drug independently developed by Suzhou Henrui Pharmaceutical Co., Ltd., which can selectively block the activation of PD-1 and its downstream signaling pathway, and restore immune function by activating effector T lymphocytes and cell-mediated immune response.Some studies have shown that the application of carrelizumab in patients with advanced solid tumors shows some clinical value, and predictive biomarkers such as PD-L1 expression level and tumor mutation load can screen out patients with high response to PD-1/PD-L1 monoclonal antibodies.Even so, PD1/PD-L1 blocking therapy provides clinical benefit in less than 20% of cancer patients，suggesting that patients using these drugs rely solely on their insufficient preexisting endogenous anti-tumor specific T cells.Anti-angiogenic drugs can specifically bind to vascular endothelial growth factor (VEGF) and its receptor 2(VEGFR2), achieving the dual effect of enhancing cytotoxic chemotherapy and achieving molecular targeted therapy.Some recent studies have shown that angiogenesis inhibitors can regulate tumor microenvironment and relieve hypoxia of tumor cells, which may promote tumor immune recovery .Ramvatinib mesylate is a class of multi-target receptor tyrosine kinase inhibitors, which can block a series of regulatory factors including VEGFR1-3, KIT and RET in tumor cells, and significantly inhibit angiogenesis in tumor tissues.It is currently FDA approved as a first-line treatment for patients with unresectable hepatocellular carcinoma.In a phase III clinical study, the overall survival of remvatinib in the first-line treatment of unresectable hepatocellular carcinoma was comparable to sorafenib (13.6 vs12.3 months) .Another basic study showed that rumvatinib modulates cancer immunity in the tumor microenvironment by reducing tumor-associated macrophages (TAM), and that when combined with PD-1 inhibitors, it can enhance anti-tumor activity through the IFN signaling pathway.In addition, previous studies have found that transarterial chemoembolization (TACE) combined with antiangiogenic agents in the treatment of advanced hepatocellular carcinoma shows a good response to tumor treatment compared with TACE alone, but the incidence of treatment-related adverse events is high and the survival time of patients is not significantly improved.Therefore, in this study, TACE, the powerful anti-angiogenic drug Ramvatinib and the new PD-1 inhibitor Carrizumab were combined to treat liver cancer patients, so as to improve the quality of life of patients and improve their survival benefits.This study aims to explore the clinical outcomes of TACE, Ramvatinib combined with carririzumab in patients with stage BCLCB/C liver cancer, monitor the complications and tumor treatment response of patients, study the appropriate population for combined treatment, and evaluate the hepatorenal and cardiotoxicity of the drugs in humans.Focusing on exploring the mechanism and application value of antiangiogenic therapy combined with immunotherapy in the treatment of liver cancer, to provide new treatment options for patients with middle and advanced liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* From 18 to 75 years old, there are no gender restrictions, and the pre-survival period exceeds 12 weeks;
* Primary liver cancer diagnosed by clinical and imaging studies, histology or cytology;
* Liver cancer patients with B/C stage according to BCLC staging;
* Have not used molecular targeted therapy drugs or immune checkpoint inhibitors in the past;
* The behavioral status score of the Eastern Cooperative Oncology Group (ECOG) is 0 or 1;
* The main organ functions are normal, and there is no serious blood, heart, lung, liver, kidney dysfunction and immune deficiency diseases. Laboratory examination meets the following requirements: a. Hemoglobin (HGB) ≥ 90g/L; b. Neutrophil count (ANC) ≥ 1.5×109/L; c. Platelet count (PLT) ≥ 100×109/L; d. ALT and AST≤2.5×ULN; liver metastasis, then ALT and AST≤5×ULN; e. total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); f. serum Cr≤1'ULN, Endogenous creatinine clearance rate>50ml/min (Cockcroft-Gault formula); g. Urine routine is normal, or urine protein <(++), or 24-hour urine protein <1.0 g;
* The coagulation function is normal, without active bleeding and thrombosis: a. International standardized ratio INR≤1.5×ULN; b. Partial thromboplastin time APTT≤1.5×ULN; c. Prothrombin time PT≤1.5×ULN ；
* The subject voluntarily joined the study and signed an informed consent form.

Exclusion Criteria:

* Suffer from active malignant tumors other than liver cancer within five years or at the same time. Cured localized tumors, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, etc. can be included in the group;
* Liver cancer tumor size ≥ 70% of liver parenchyma or extrahepatic metastasis;
* Pregnant or lactating women;
* Known allergy to carrelizumab, lenvatinib or pharmaceutical excipients;
* Go through other anti-tumor treatments, including surgical treatment, local treatment and systemic treatment within 4 weeks before enrollment;
* Have received organ or allogeneic bone marrow transplantation;
* Suffer from any active autoimmune disease or history of autoimmune disease (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, thyroid ·Reduced function (can be included after hormone replacement therapy)); Immune suppressive drugs have been used within 14 days before the first use of the study drug, excluding nasal spray and inhaled corticosteroids or physiological doses of systemic steroid hormones (ie not more than 10 mg/day prednisolone or equivalent drug physiology Doses of other corticosteroids);
* Vaccination of live attenuated vaccine within 4 weeks before the first administration or planned during the study period;
* Severe infections (such as intravenous infusion of antibiotics, antifungal or antiviral drugs) within 4 weeks before the first administration, or unexplained fever >38.5°C during the screening period/before the first administration;
* Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* There is objective evidence showing that he has suffered from pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia, severely impaired lung function, etc.;
* Suffering from hypertension who cannot fall to the normal range after 3 months of treatment with antihypertensive drugs (systolic blood pressure ≤ 140 mmHg / diastolic blood pressure ≤ 90 mmHg);
* Suffer from uncontrollable clinical symptoms or diseases of the heart, including but not limited to congestive heart failure (NYHA grade> Ⅱ grade); unstable or severe angina pectoris; acute myocardial infarction within 6 months; clinically significant Patients with supraventricular or ventricular arrhythmia requiring clinical intervention; left ventricular ejection fraction (LVEF) <50%; Patients with active bleeding due to various reasons or patients at risk of severe bleeding, including but not limited to severe bleeding (bleeding> 30 ml within 3 months), hemoptysis (bleeding> 5 ml within 4 weeks) and occurring within 12 months Thromboembolic events (including stroke events and/or transient ischemic attacks);
* Participated in other clinical trials or participated in any other drug clinical research within 4 weeks, or no more than 5 half-lives from the last study drug;
* Other situations deemed unsuitable by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
PFS | The period of time between the date of randomization until the date of first documented progression , assessed up to 24 months
  progression free survival

SECONDARY OUTCOMES:
OS | From date of randomization until the date of death from any cause, assessed up to 24 months
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT04909866/Prot_000.pdf